CLINICAL TRIAL: NCT07231016
Title: The Protective Effect of Influenza Vaccine for Vulnerable Population
Brief Title: Influenza Vaccination Against Infectious Complications and Mortality in Older Adults With Fractures: a Large-scale Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TMU-JIRB-201910032; TMU-Joint Institutional Review (Other: TMU-Joint Institutional Review Board)
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2019-10

CONDITIONS: Fracture; Influenza Vaccination
Keywords: Influenza vaccination; infectious diseases; mortality; fracture
MeSH Terms: conditions — Fractures, Bone; Influenza, Human; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with fracture hospitalization: A retrospective cohort study was conducted utilizing data from a health insurance database in Taiwan. The study included 561,566 individuals aged 65 years and older who were hospitalized for fractures between 2009 and 2020.

SUMMARY:
Background: Both influenza and bone fractures are significant contributors to morbidity and mortality among older adults. This study evaluated the associations between influenza vaccination (IV) and adverse outcomes following fracture-related hospitalizations in elderly individuals.

Methods: A retrospective cohort study was conducted utilizing data from a health insurance database in Taiwan. The study included 561,566 individuals aged 65 years and older who were hospitalized for fractures between 2009 and 2020. Patients were stratified according to whether they had received an IV within the 12 months preceding their fracture event. Propensity score matching was employed between the vaccinated and unvaccinated groups. Multivariate logistic regression models were used to estimate adjusted odds ratios (ORs) and 95% confidence intervals (CIs) for postfracture infectious complications and 30-day mortality associated with prior IV.

DETAILED DESCRIPTION:
A nested retrospective cohort design was adopted to evaluate the influence of IVs on clinical outcomes following fracture-related hospitalizations. The analysis drew upon a nationwide, dynamic cohort comprising more than 23 million insured individuals. From this population, we identified 561,566 patients aged 65 years and older who were admitted for fracture treatment between 2009 and 2020. Among them, 213,381 individuals had received an IV within the 12 months prior to admission, whereas 348,185 had not.

To mitigate potential confounding, we applied 1:1 propensity score matching, pairing each vaccinated patient with a nonvaccinated counterpart. The matching criteria included demographic characteristics (age, sex), socioeconomic status (low-income designation), fracture type, comorbidities (documented within the previous 24 months), emergency department visits, and hospital admissions during the 12 months preceding the fracture event.

The primary outcomes were assessed within 30 days postadmission and included the occurrence of pneumonia, septicemia, urinary tract infections, intensive care, hospital length of stay, total medical expenditure, and 30-day mortality. Postfracture infectious complications were identified through physician-coded diagnoses during the index hospitalization or in subsequent inpatient and outpatient claims within 30 days. To avoid confounding due to preexisting infections, individuals with documented cases of pneumonia or septicemia within the six months before fractures were excluded from the analysis.

ELIGIBILITY:
Inclusion Criteria:

Patients with fracture hospitalization who aged more than 65 years

Exclusion Criteria:

People had no fracture hospitalization and people aged lower than 65 years

Min Age: 20 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study utilized a nationwide, population-based cohort encompassing over twenty million insured individuals. From this cohort, we identified older adults admitted for fracture treatment between 2009 and 2020. Among them, approximately two in five had received an influenza vaccination within the year before hospitalization. To minimize confounding, we performed one-to-one propensity score matching, pairing each vaccinated patient with an unvaccinated counterpart based on demographic, socioeconomic, and clinical characteristics, including age, sex, income status, fracture type, comorbidities, and prior healthcare utilization.
Sampling Method: Probability Sample
Enrollment: 561566 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
post-fracture 30-day mortality | 30-day period after fracture hospitalization
  We calculated the mortality after fracture hospitalization within 30-day period.
mortality after fracture | 30-day period after fracture hospitalization
  30-day mortality after fracture hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chang Liao, PhD, MPH, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT07231016/Prot_SAP_000.pdf